CLINICAL TRIAL: NCT03635125
Title: A Prospective, Randomized, Open-Label, Active-Comparator, Blinded-Endpoint, 12-week Forced-Titration Study of the Efficacy and Safety of Nebivolol Verses Metoprolol in Hypertensive Subjects Taking Amlodipine
Brief Title: Efficacy and Safety of Nebivolol Versus Metoprolol in Hypertensive Subject Taking Amlodipine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trinity Hypertension & Metabolic Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BYS-MD-48
Record Dates: First submitted 2018-03-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: JNC 7 Stage 1 or 2 Hypertension

STUDY DESIGN:
Intervention Model Description: 12-week Amlodipine background treatment phase followed by a 4-week Low dose Nebivolol/Metoprolol treatment phase and a 4-week high dose Nebivolol/Metoprolol treatment phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Background treatment phase (No Intervention): A 12- week Amlodipine 10 mg background treatment phase
- Low Dose Treatment Phase-Nebivolol I (Active Comparator): 4-week low dose Nebivolol10 mg/Metoprolol 50 mg treatment phase
  Interventions: Drug: Nebivolol I; Drug: Nebivolol II
- High dose treatment Phase-Nebivolol II (Active Comparator): 4-week High dose Nebivolol 20 mg/Metoprolol 100mg treatment phase
  Interventions: Drug: Nebivolol I; Drug: Nebivolol II
- Baseline Washout Phase (Other): 2 to 4 week Baseline Washout Phase
  Interventions: Other: Baseline Washout Phase

INTERVENTIONS:
Drug: Nebivolol I — Low dose treatment phase: Nebivolol 10 mg or Metoprolol 50 mg High dose treatment phase: Nebivolol 20 mg or Metoprolol 100mg
  Other Names: Metoprolol I
  Arms: High dose treatment Phase-Nebivolol II; Low Dose Treatment Phase-Nebivolol I
Drug: Nebivolol II — Low dose treatment phase: Nebivolol 10 mg or Metoprolol 50 mg High dose treatment phase: Nebivolol 20mg or Metoprolol 100mg
  Other Names: Metoprolol II
  Arms: High dose treatment Phase-Nebivolol II; Low Dose Treatment Phase-Nebivolol I
Other: Baseline Washout Phase — 2 to 4 week Baseline Washout Phase
  Arms: Baseline Washout Phase

SUMMARY:
Study is to evaluate the effect of Nebivolol to treat high blood pressure compared to an already approved drug, Metoprolol ER with background treatment of Amlodipine.

DETAILED DESCRIPTION:
Open-label, single center study consisting of a 2 to 4 week baseline washout phase, a 12-week Amlodipine background treatment phase followed by a 4-week Low Dose Nebivolol/Metoprolol Treatment phase and a 4-week High Dose Nebivolol/Metoprolol Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Capable of reading, comprehending the consent process and providing written informed consent to participate in the study.
* Male or female equal/over 18 years of age.
* Stage I-II hypertension defined as a baseline mean seated cuff Diastolic blood pressure of equal/over 95 mmHg and equal/less 115 mmHg and Systolic blood pressure equal/less to 180 mmHg at two consecutive qualifying visits during the placebo run in period.
* Arm circumference less 45 cm
* Compliance with single blind placebo capsules between V1-4 of 80-120%.
* Women may be enrolled if all three of the following criteria are met:
* Have a negative serum pregnancy test at screening
* Are not breastfeeding
* Do not plan to become pregnant during the study and if one of the three criteria is met:
* Have had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form
* Have been postmenopausal for at least 1 year
* Are of childbearing potential and will practice one the following methods of birth control throughout the study: oral, patch, injectable, or implantable hormone contraception, intrauterine device, diaphragm plus spermicide or female condom plus spermicide. Abstinence, partner's vasectomy are not acceptable methods of contraception.

Exclusion Criteria:

* Known allergy or hypersensitivity to Beta Blockers.
* Known allergy or hypersensitivity to Calcium Channel Blockers.
* Patients with severe hypertension (mean seated cuff Diastolic blood pressure > 115 mmHg or mean seated Systolic blood pressure >180 mmHg) or any form of secondary hypertension.
* Patients within the past 6 months with a history of hypertensive encephalopathy, stroke or transient ischemic attack.
* Patients within the last 6 months with a history of myocardial infarction, percutaneous trans luminal coronary revascularization, coronary bypass graft, valvular surgery or unstable angina.
* Patients with evidence of resting bradycardia (<50 bpm) via palpation.
* Patients with a history of heart block greater than First Degree Sino atrial Block. Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial Fibrillation, Atrial Flutter, Congestive Heart Failure, or other manifestations of clinically significant cardiac valvular disease.
* Patients with hemodynamically significant cardiac valvular disease.
* Patients with evidence of significant chronic renal impairment as indicated by a serum creatinine of > 2.5mg/dL
* Patients with evidence of liver disease as indicated by AST (SGOT) or ALT (SGPT) > 2.5 times or total bilirubin > 1.5 times, the upper limit of the laboratory normal range.
* Patients who demonstrate other laboratory test values deviating from the Normal range which are considered to be clinically significant by the investigator.
* Patient with a history or presence of gastrointestinal disease which may interfere with drug absorption.
* Patients with insulin and non-insulin dependent diabetes mellitus not controlled on diet, insulin or oral hypoglycemic as defined by a HgA1c >10.
* Severe psychological or emotional condition which may interfere with participation in the study.
* History of or current use of illicit drugs or alcohol abuse.
* Participation in a clinical trial and taking any investigation drug within 30 days prior to enrolling into the study (Screening Visit).
* A physical condition that would limit accurate BP measurement.
* Inability to swallow a tablet or capsule.
* History of moderate or sever asthma or Chronic obstructive pulmonary disease.
* Any other medical condition which, in the Investigator's opinion, may render the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08-30 (Actual); Primary Completion 2011-05-26 (Actual); Study Completion 2011-07-18 (Actual)

PRIMARY OUTCOMES:
Mean Change from baseline in trough Diastolic Blood Pressure | 4 and 8 weeks of treatment
  Mean change by millimeters of mercury from baseline in trough Diastolic Blood Pressure
Mean Change in Edema Measurement | 4 and 8 weeks of treatment
  Mean change in edema measurement by water immersion of treatment in millimeters of water

SECONDARY OUTCOMES:
Change from baseline in trough Systolic blood pressure of treatment. | 4 and 8 weeks of treatment
  Change from baseline by millimeters of mercury in trough Systolic blood pressure of treatment.
Percentage of subjects achieving Blood pressure goals | 4 and 8 weeks of treatment
  Percentage of subjects achieving Blood pressure goals of either Nebivolol compared to Metoprolol

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Punzi, MD, Principal Investigator — Punzi Medical Center
Locations (1):
- Punzi Medical Center, Carrollton, Texas, United States

IPD SHARING:
Plan to Share IPD: No